CLINICAL TRIAL: NCT02522026
Title: Follow-up-study of Participants (COPD Patients and Healthy Control Subjects) From the Cross-sectional Study "11-03 Ribolution" for the Evaluation of Predictive Biomarkers Based on Non-coding RNA
Brief Title: Follow-up-study of COPD Patients and Healthy Controls for Evaluation of Predictive Non-coding RNA Biomarkers
Acronym: Ribo2
Status: Completed | Type: Observational
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jens Hohlfeld, MD, Division Director Airway Research, Fraunhofer-Institute of Toxicology and Experimental Medicine
Other Study IDs: 15-01 RIBO II
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy volunteers
- Healthy smokers
- COPD GOLD1
- COPD GOLD2
- COPD GOLD3/4

SUMMARY:
Between 2012 and 2014, a cohort of 90 COPD subjects of disease severity grades GOLD I-IV as well as 60 healthy control subjects (30 smokers and 30 non-smokers) have been examined regarding different clinical and blood/ sputum derived biomarkers at the investigators' research center. This observation study will follow-up/re-examine all available subjects regarding disease course and treatment changes after 3 years (+/-6 months) for the investigation of ncRNA/ transcriptome biomarkers for their potential to indicate disease progression. In addition, biobanking of respective biosamples for potential future COPD biomarker research will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Study "11-03 Ribolution"
* Able and willing to give written informed consent
* Not pregnant, as confirmed by pregnancy test

Exclusion Criteria:

* Past or present disease occurred since participation in "11-03 Ribolution", which as judged by the investigator, may affect the outcome of the study.
* Serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study or impact on subject safety
* Has experienced a significant upper or lower respiratory tract infection incl. moderate or severe exacerbation (requiring oral corticosteroid, antibiotics or hospitalisation) within the last 4 weeks. All courses of oral corticosteroids and antibiotics must be completed at least 4 weeks before study start
* Clinically significant pathological findings in safety laboratory tests having an impact on study participation.
* Actual drug or alcohol abuse.
* Suspected inability to understand and follow protocol requirements, instructions, study-related restrictions, and to understand nature, scope, and possible consequences of the study.
* Being a vulnerable subject (dependent, in detention, or without mental capacity)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All 150 patients of study "11-03 Ribolution" will be contacted and re-invited for the current follow-up study as completely as possible
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Lung volumes by pulmonary function testing | after 3 years ± 6 months
  forced expiratory volume in 1 second

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Hohlfeld, Prof, Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine
Locations (1):
- Fraunhofer-Institute for Toxicology and Experimental Medicine, Hanover, Germany